CLINICAL TRIAL: NCT02494713
Title: Neoadjuvant Androgen Deprivation Therapy and Chemotherapy Followed by Radical Prostatectomy in Patients With Prostate Cancer
Brief Title: Hormonal Therapy and Chemotherapy Followed by Prostatectomy in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment; resource re-allocation
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robert J Amato, Professor and Director, Division of Oncology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-14-101; HSC-MS-14-0424 (Other: UTHSC-H CPHS (IRB))
Record Dates: First submitted 2015-06-23; First posted 2015-07-10 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: Advanced Prostate Cancer; Neoadjuvant; Hormone therapy; ADT; Androgen Deprivation Therapy; Chemotherapy; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Doxorubicin; Ketoconazole; Docetaxel; Estramustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADT + chemotherapy (Other): Patients will be treated with 4 monthly injections of degarelix along with two 8-week cycles of chemotherapy (doxorubicin and ketoconazole, weeks 1, 3, 5 and docetaxel and estramustine, weeks 2, 4, 6). Each cycle of chemotherapy will consist of 6 weeks of chemotherapy and 2 weeks of rest. In the absence of toxicity or disease progression, patients will receive 2 cycles of treatment prior to radical prostatectomy.
  Interventions: Drug: Degarelix; Drug: Doxorubicin; Drug: Ketoconazole; Drug: Docetaxel; Drug: Estramustine

INTERVENTIONS:
Drug: Degarelix — Subcutaneous injection, once/month for 4 months
  Other Names: Firmagon; degarelix acetate
Drug: Doxorubicin — 20 mg/m2 as a 24-hour intravenous infusion on day 1 each week, weeks 1, 3, and 5
  Other Names: Adriamycin
Drug: Ketoconazole — 400 mg orally 3 times daily for 7 days, in weeks 1, 3, and 5
  Other Names: Nizoral
Drug: Docetaxel — 35 mg/m2 intravenously on day 1 of each week, weeks 2, 4, and 6
  Other Names: Taxotere
Drug: Estramustine — 280 mg orally 3 times daily for 7 days, in weeks 2, 4, and 6
  Other Names: Emcyt

SUMMARY:
This is a study for men who have locally-advanced prostate cancer and are eligible to undergo prostatectomy. Standard treatment is prostatectomy alone, but there is a chance that cancer may spread to other organs in the future, even after the prostate is removed. If this were to occur, standard treatment would be androgen deprivation therapy (ADT; hormone therapy that blocks testosterone) plus chemotherapy. Clinical trials suggest that neoadjuvant treatment (treatment given before primary therapy) may prevent a recurrence. The purpose of this research study is to assess the safety and benefit of ADT plus chemotherapy given before prostate removal.

DETAILED DESCRIPTION:
This is an open-label, single-arm study of neoadjuvant ADT and chemotherapy in subjects with non-metastatic, locally-advanced prostate cancer who are eligible for radical prostatectomy.

Patients will be treated with 4 monthly injections of degarelix along with two 8-week cycles of chemotherapy. Each cycle of chemotherapy will consist of 6 weeks of chemotherapy and 2 weeks of rest. In the absence of toxicity or disease progression, patients will receive 2 cycles of treatment prior to radical prostatectomy.

The primary endpoint will be complete or near-complete pathologic response.

Safety will be assessed on any patient receiving at least one dose of study drug by the reporting of adverse events, vital signs and by the assessment of findings on physical exam and routine safety laboratory determinations. The severity of adverse events and certain abnormal laboratory findings will be assessed according to the NCI CTCAE V4.03.

Laboratory-based studies will evaluate the following:

* Complete metabolic profile

  o BUN, creatinine, alkaline phosphatase, ALT/AST, total bilirubin, LDH, calcium, albumin, glucose, magnesium, uric acid, phosphorous
* Electrolytes

  o Sodium, potassium, chloride, CO2 content
* Hematology

  * CBC with differential, platelet count
  * PT, INR, PTT
* Testosterone
* Biomarkers

  * PSA
  * CTCs

ELIGIBILITY:
Inclusion Criteria:

* Pathologic proof of prostatic adenocarcinoma without evidence of regional and/or distant metastasis, clinical stage T1c or T2a with high grade disease (Gleason 8-10) on initial biopsy, clinical stage T2b-T2c with Gleason grade 7 (4+3), or clinical stage T3. No neuroendocrine differentiation or small cell features.
* Recent (<6 weeks prior to study entry) negative bone scan and CT of the chest and abdomen.
* Appropriate surgical candidate for radical prostatectomy and a performance status of <2 (ECOG scale).
* Adequate bone marrow function as defined as an absolute peripheral granulocyte count >1500 and platelet count >100,000.
* Adequate hepatic function per the following criteria:

  * Albumin ≥2.8 g/dL
  * AST and ALT ≤5 x ULN
  * Total bilirubin <2 mg/dL
* Adequate renal function per the following criteria:

  o Serum creatinine ≤1.5 x ULN
* Normal coagulation profile (INR ≤ 1.5, aPTT ≤ 1.5 x ULN for the lab) and no history of substantial non-iatrogenic bleeding diatheses. Use of anticoagulants is limited to local use only (for control of central line patency).
* Age ≥ 18 years
* Written informed consent to participate in this study.

Exclusion Criteria:

* Prostatic adenocarcinoma with neuroendocrine differentiation or small cell features
* Surgical resection or major surgery within 4 weeks or stereotactic biopsy within 1 week of first ADT and chemotherapy treatment
* Previous or current hormonal treatment, chemotherapy, radiation therapy, immunotherapy, or investigational study drug.
* Unable to tolerate multiparametric MRI or is contraindicated.
* Patients not appropriate surgical candidates for radical prostatectomy based on the evaluation of coexistent medical diseases and competing causes of death.
* Patients with uncontrolled cardiac, hepatic, renal, or neurologic/psychiatric disorder.
* Severe gastrointestinal bleeding within 12 weeks of treatment with ADT and chemotherapy
* Patients who are HIV positive or have chronic hepatitis B or C infections.
* Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, unless a 2D echocardiogram or multi-gated acquisition scan (MUGA) performed within 3 months of enrollment demonstrates a left ventricular ejection fraction >45%.
* Sensory neuropathy grade >1.
* History of another malignancy within the previous 5 years other than curatively treated non-melanoma skin cancer.
* Use of herbal products that may decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within 4 weeks of enrollment.
* Any other condition, including concurrent medical condition, social circumstance or drug dependency, which in the opinion of the investigator could compromise patient safety and/or compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, D.O., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth Memorial Hermann Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADT + Chemotherapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 58 [49 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status scale measures level of functioning. The scale ranges from 0 to 5, with 0 indicating the highest level of functioning and 5 the lowest.
  Participants
    0 | 4
    1 | 0
    2 | 0
    3 | 0
    4 | 0
    5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Measured by Pathologic Response
Description: Pathologic response is defined by percentage of tumor burden remaining at time of prostate removal. Percentage of tumor burden is measured based on a pathologist's assessment of the prostate tissue removed and visual estimate of how much tumor there is in the prostate.
Time Frame: Day of prostate removal, which is about 5 months following the day participant signed consent.
Measure: Median (Full Range); unit: percentage of tumor burden remaining
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
percentage of tumor burden remaining | 30 [1 to 70]

2. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: Prostate-specific antigen, or PSA, is a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis. The results are reported as nanograms of PSA per milliliter (ng/mL) of blood.
Time Frame: baseline
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
ng/mL | 58.7 [44.7 to 77.4]

3. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: as for outcome 2
Time Frame: Cycle 2 Day 1, about 8 weeks after treatment initiation (but before prostatectomy)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
ng/mL | 0.4 [0.1 to 2.9]

4. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: as for outcome 2
Time Frame: Cycle 2 Day 57, about 16 weeks after treatment initiation (but before prostatectomy)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
ng/mL | 0.15 [0.01 to 2]

5. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: as for outcome 2
Time Frame: Day 133, about 19 weeks after treatment initiation (but before prostatectomy)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
ng/mL | 0.055 [0.01 to 1.3]

6. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: as for outcome 2
Time Frame: about 20 weeks after treatment initiation (day of prostatectomy)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
ng/mL | 0.01 [0.01 to 0.1]

7. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: as for outcome 2
Time Frame: about 32 weeks after treatment initiation (about 12 weeks after prostatectomy)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
ng/mL | 0.01 [0.01 to 0.1]

8. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: as for outcome 2
Time Frame: about 44 weeks after treatment initiation (about 24 weeks after prostatectomy)
Population: This data was only collected for 3 out of the 4 participants.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 3
ng/mL | 0.35 [0.2 to 0.5]

9. Secondary Outcome: Efficacy as Measured by Prostate-specific Antigen (PSA) Levels
Description: as for outcome 2
Time Frame: about 68 weeks after treatment initiation (about 48 weeks after prostatectomy)
Population: This data was collected for only 3 out of the 4 participants.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 3
ng/mL | 0.1 [0.01 to 0.8]

10. Secondary Outcome: Efficacy as Measured by Circulating Tumor Cell (CTC) Numbers
Time Frame: From the time the participant signs the informed consent until prostatectomy, an average of 5 months.
Population: This data was not collected for any participants.
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 0

11. Secondary Outcome: Efficacy as Measured by Volume of the Prostate Tumor as Assessed by Multiparametric Prostate Magnetic Resonance Imaging (mpMRI)
Description: The volume of the prostate tumor was measured by a radiologist's assessment of multiparametric prostate magnetic resonance imaging.
Time Frame: baseline
Measure: Median (Full Range); unit: cc
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
cc | 19.3 [13.3 to 26.1]

12. Secondary Outcome: Efficacy as Measured by Volume of the Prostate Tumor as Assessed by Multiparametric Prostate Magnetic Resonance Imaging (mpMRI)
Description: as for outcome 11
Time Frame: post treatment but prior to prostatectomy (about 25 days after the end of treatment)
Measure: Median (Full Range); unit: cc
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
cc | 3.75 [1.3 to 7.4]

13. Secondary Outcome: Safety of Drug Regimen as Measured by Number of Adverse Events
Description: Number of adverse events was measured as a count of all participant adverse events that occurred from the time participant first initiates ADT plus chemotherapy until participant's completion of neoadjuvant ADT plus chemotherapy.
Time Frame: From the time participant first initiates ADT plus chemotherapy until participant's completion of neoadjuvant ADT plus chemotherapy.
Measure: Number; unit: adverse event
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
adverse event | 119

14. Secondary Outcome: Surgical Morbidity as Measured by Number of Adverse Events
Description: Number of adverse events was measured as a count of all participant adverse events that occurred from the time participant first initiates ADT plus chemotherapy until the participant was taken off-study or the study was stopped, an average of 20 months
Time Frame: From the time the participant signs the informed consent until the participant was taken off-study or the study was stopped, an average of 20 months
Measure: Number; unit: adverse event
Arm/Group | ADT + Chemotherapy
Number analyzed (Participants) | 4
adverse event | 119

ADVERSE EVENTS:
Time Frame: From the time the participant signs the informed consent until the participant was taken off-study or the study was stopped, an average of 20 months.
Arm/Group | ADT + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADT + Chemotherapy (N=4)
WATERY EYES (Eye disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 2 (6)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 2 (4)
DRY MOUTH (Gastrointestinal disorders) | 1 (2)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 2 (9)
NAUSEA (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
BACK PAIN (General disorders) | 1 (2)
EDEMA LIMBS (General disorders) | 3 (9)
FATIGUE (General disorders) | 4 (12)
FLU LIKE SYMPTOM-ACHINESS (General disorders) | 1 (1)
INJECTION SITE REACTION (General disorders) | 2 (3)
MALAISE (General disorders) | 1 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PAIN (General disorders) | 2 (3)
INFECTIONS/INFESTATIONS, THRUSH (Infections and infestations) | 1 (1)
BRUISING - PORT A CATH SITE (Injury, poisoning and procedural complications) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (6)
MUSCULOSKELETAL/CONNECTIVE TISSUE DISORDERS, MUSCLE ACHES (Musculoskeletal and connective tissue disorders) | 1 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 2 (4)
HEADACHE (Nervous system disorders) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 2 (5)
PSYCHIATRIC DISORDER, EMOTIONAL (Psychiatric disorders) | 1 (2)
RESTLESSNESS (Psychiatric disorders) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 2 (3)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (4)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN/SQ TISSUE DISORDERS, PEELING OF SKIN AT PORT A CATH SITE (Skin and subcutaneous tissue disorders) | 1 (1)
FLUSHING (Vascular disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 2 (2)
PSYCHIATRIC DISORDER, ANGER (Psychiatric disorders) | 1 (1)
SKIN/SQ TISSUE DISORDERS, RIGHT HAND SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed and limited data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT02494713/Prot_SAP_000.pdf